CLINICAL TRIAL: NCT00229164
Title: The Effect of Transcutaneous Electric Nerve Stimulation on Primary Dysmenorrhea-a Randomized Control Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 9361701148
Record Dates: First submitted 2005-09-27; First posted 2005-09-29 (Estimated); Last update posted 2012-12-27 (Estimated); Status verified 2012-11

CONDITIONS: Primary Dysmenorrhea,
Keywords: Primary Dysmenorrhea,; Transcutaneous Electric Nerve Stimulation
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Transcutaneous Electric Nerve Stimulation (TENS)

SUMMARY:
The purpose of this study is to investigate the effect of high frequency TENS and compare to the placebo effect by sham TENS in a randomized control study.

DETAILED DESCRIPTION:
Over 50% of American women suffered from dysmenorrhea and 10% of them will take sick leave for 1-2 days. Previous randomized control studies have demonstrated the pain relief effect of using high frequency TENS in dysmenorrheal pain. However, no investigation has been conducted to investigate the effect of high frequency TENS in female population in our country. The purpose of this study is to investigate the effect of high frequency TENS and compare to the placebo effect by sham TENS in a randomized control study.

ELIGIBILITY:
Inclusion Criteria:

* primary Dysmenorrhea

Exclusion Criteria:

* subjects with organic disorders

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2005-10; Study Completion 2006-01

PRIMARY OUTCOMES:
all measure the pain threshold,
self-rating questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Shwu-Fen Wang, Ph.D, Study Director — School and Graduate Institute of Physical Therapy, College of Medicine, National Taiwan University